CLINICAL TRIAL: NCT01742429
Title: Levoﬂoxacin and Bismuth-containing Therapy Versus Quadruple Therapy as Second-line Treatment of Resistant Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Prof. of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2012008
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2013-06

CONDITIONS: Cure Rate of Helicobacter Pylori Infection
Keywords: Helicobacter pylori; second line treatment
MeSH Terms: interventions — Proton Pump Inhibitors; bismuth subsalicylate; Metronidazole; Tetracycline; Amoxicillin; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levofloxacin-bismuth therapy (Experimental): 14 day levoﬂoxacin and bismuth-containing therapy:PPI,bismuth, amoxicillin, levoﬂoxacin
  Interventions: Drug: Proton pump inhibitor; Drug: Bismuth subsalicylate; Drug: Amoxicillin; Drug: Levofloxacin
- classical quadruple therapy (Active Comparator): 14 day classical quadruple therapy:PPI,bismuth, metronidazole, tetracycline
  Interventions: Drug: Proton pump inhibitor; Drug: Bismuth subsalicylate; Drug: Metronidazole; Drug: Tetracycline

INTERVENTIONS:
Drug: Proton pump inhibitor
Drug: Bismuth subsalicylate
Drug: Metronidazole — antibiotic
  Arms: classical quadruple therapy
Drug: Tetracycline — antibiotic
  Arms: classical quadruple therapy
Drug: Amoxicillin — antibiotic
  Arms: Levofloxacin-bismuth therapy
Drug: Levofloxacin — antibiotic
  Arms: Levofloxacin-bismuth therapy

SUMMARY:
To test the efﬁcacy of 14 day levoﬂoxacin and bismuth-containing second-line therapy for resistant Helicobacter pylori infection, to compare with the classical quadruple therapy.

ELIGIBILITY:
Inclusion Criteria:

* all patients had failed H.pylori therapies including clarithromycin, metronidazole and/or amoxicillin (if not allergic) before.

Exclusion Criteria:

* patients less than 18 years old,
* previous gastric surgery,
* pregnancy,
* lactation,
* major systemic diseases,
* administration of antibiotics,
* bismuth,
* antisecretory drugs in the preceding 8 weeks, or
* allergy to any one of the medication used in the quadruple regimens.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
eradication rate | 2 months
  urease breath test

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China